CLINICAL TRIAL: NCT04558580
Title: A Double-Blind, Placebo-Controlled, Parallel-Group Study of Rufinamide Given as Adjunctive Therapy in Patients With Refractory Partial Seizures
Brief Title: Safety Study of Rufinamide Given as an add-on Therapy to Treat Patients With Seizures
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2080-A001-301
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Refractory Partial Seizures
Keywords: Seizure, Seizures, Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — rufinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention)
- Rufinamide (Experimental)
  Interventions: Drug: Rufinamide

INTERVENTIONS:
Drug: Rufinamide — Rufinamide
  Arms: Rufinamide

SUMMARY:
This study will evaluate the efficacy and safety of Rufinamide in reducing seizure frequency in subjects with partial seizures not fully controlled despite treatment with 1 to 3 concomitant antiepileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients between 12 and 80 years of age
* Dx of epilepsy with partial onset seizures woth or woth out secondarily generalized seizures
* Non controlled partial seizures despite treatment with 2 different AEDs for at least 2 years
* must have 6 seizures during baseline
* current treatment with maximum of 3 AEDs
* stable dose of AED(s)for at least 1 month
* if patient has VNS, must have been implanted 6 months prior to randomization

Exclusion Criteria:

* Participation in any investigational product for at least 1 month prior to visit 1
* Presence of non-motor simple partial seizures only
* presence of generalized epilepsies
* Evidence of clinically significant disease
* Clinically significant ECG
* Psychogenic seizure in previous year
* History of drug/alcohol abuse
* History of suicide attempt
* Multiple drug allergies
* Concomitant felbamate use
* Need for frequent rescue benzodiazepines
* Concomitant use of vigabatrin
* All patients diagnosed with congenital short QT syndrome

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Percentage change in total partial seizure frequency from baseline. | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Maertens, MD, Principal Investigator — University of South Alabama
Locations (1):
- University of South Alabama, Mobile, Alabama, United States